CLINICAL TRIAL: NCT04522518
Title: To Hear Diverse Voices: Self-identified Participation Goals and Environmental Supports and Barriers of Children With Disabilities
Brief Title: Self-identified Participation and Environment of Children With Disabilities
Status: Completed | Type: Observational
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Lin-Ju Kang, Associate Professor, Chang Gung University
Other Study IDs: 201812ES010
Record Dates: First submitted 2020-08-12; First posted 2020-08-21 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Developmental Disability
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DD group: 160 pairs of children with disabilities 6-12 years of age and their caregivers (n=320)
  Interventions: Device: PmP-C App
- TD group: 160 pairs of typically developing children 6-12 years of age and their caregivers (n=320)
  Interventions: Device: PmP-C App

INTERVENTIONS:
Device: PmP-C App — The key features of PmP-C App include: "About Me" (entering child's demographic data e.g. age, gender, family members), "My participation" (answering frequency and involvement of activities), and "My goal" (selecting 3 important activities they desire to change and identify things that made them easy or hard to do, i.e. participation goals and environmental supports or barriers). The App is to be manipulated adult interviewers but also can be manipulated by the child if they are able to.

SUMMARY:
Picture My Participation (PmP) is a child self-report tool for children and adolescents with disabilities. The PmP uses pictures that enable children to identify participation frequencies, participation goals, and environmental supports/barriers to a home, school, and community activities. The PmP has been translated to different languages and cultures, including Traditional Chinese for the use in Taiwan. Given the advances and popularity of mobile technologies, the PmP-Traditional Chinese version has been developed into App software (PmP-C App) to provide a fun and user-friendly interface to promote communication and active engagement in the assessment process. The PmP-C App version would be need to establish the usability, reliability and validity in children with various types of disabilities.

The purposes of this study are to: establish usability, reliability, and validity using the PMP App version, and characterize child-identified participation goals and identify environmental supports and barriers in children with and without disabilities. Data will be collected by examination and interviews using the PmP-C App and other measures for validation.

DETAILED DESCRIPTION:
This is a two-year cross-sectional study to explore the use of the PmP-C App version with children with and without disabilities. The estimated participants are 160 pairs of children with disabilities 6-12 years of age and their caregivers and 160 age-matched peers with typical development and their caregivers (a total of 640 participants). The design enables validation of the responses of children with disabilities with various sources (i.e. caregivers' responses, children without disabilities, and other child-report measures). Findings of reliability and validity will provide a basis for reporting child-identified participation goals and environmental factors. The COnsensus-based Standards for the selection of health Measurement Instruments (COSMIN) guideline is used to design a high-quality validation study. To characterize child-perceived participation and environment, the data are collected for two groups: one group of children with disabilities (the DD group) and one group of children without disabilities (the TD group). The design enables examination of how prioritized activities and frequent encountered environmental supports and barriers may vary given different capabilities of children with disabilities and peers with typical development.

ELIGIBILITY:
Children with disabilities

Inclusion Criteria:

* children aged 6 to 12 years old
* children with an identified disability or health conditions through early intervention or Disability Evaluation System in Taiwan
* children have a cognitive level of at least 5 years developmental age in receptive language based on the Peabody Picture Vocabulary Test-Revised (PPVT-R) test
* children are able to make choices between 4 options (tested by three trial questions) and are able to express their thoughts verbally, in writing/typing, or with Augmentative and Alternative Communication (AAC)
* both the child and caregiver agree to join this study

Exclusion Criteria:

* children with unstable health conditions, such as cancer, having surgery within 3 months, infection, or other active medical conditions that affect their recent daily lives
* children with progressive disease (e.g. neuromuscular disease) or degenerative disorders (e.g. degenerative seizures)
* children who are non-communicable, with uncorrected vision or hearing impairments that cannot see the instruments or hear the interview questions
* children and/or caregivers who do not understand Chinese well and thus cannot complete the instruments

Children with typical development

Inclusion criteria:

* children aged 6 to 12 years old
* children without identified disability, physical or mental health conditions related to developmental disabilities
* children are able to make choices between 4 options (tested by three trial questions) and are able to express their thoughts verbally
* both the child and caregiver agree to participate in this study

Exclusion criteria:

* children with unstable health or medical conditions (e.g. trauma or infection)
* children and/or caregivers who do not understand Chinese well and thus cannot complete the instruments

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with disabilities 6-12 years old and their parents or primary caregivers; age-matched children with typical development and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Traditional Chinese version of Picture my Participation (PmP-C) frequency scores | day 1
  The PmP-C participation frequency is scored on a 4-point scale (1=never to 4=always), a higher score indicating the higher frequency of attending in an activity.
Traditional Chinese version of Picture my Participation (PmP-C) frequency scores | 1 week since day 1 for test-retest reliability
  The PmP-C participation frequency is scored on a 4-point scale (1=never to 4=always), a higher score indicating the higher frequency of attending in an activity.
Traditional Chinese version of Picture my Participation (PmP-C) involvement scores | day 1
  The PmP-C level of involvement is scored on a 3-point scale (1= minimally involved to 3= very involved), a higher score indicating the higher perceived level of involvement when attending an activity.
Traditional Chinese version of Picture my Participation (PmP-C) involvement scores | 1 week since day 1 for test-retest reliability
  The PmP-C level of involvement is scored on a 3-point scale (1= minimally involved to 3= very involved), a higher score indicating the higher perceived level of involvement when attending an activity.
Traditional Chinese version of Picture my Participation (PmP-C) important activities | day 1
  The participants select up to 3 important activities among the PmP-C items, the item numbers will be reported.
Traditional Chinese version of Picture my Participation (PmP-C) important activities | 1 week since day 1 for test-retest reliability
  The participants select up to 3 important activities among the PmP-C items, the item numbers will be reported.

SECONDARY OUTCOMES:
Perceived Efficacy and Goal Setting (PEGS) scores | day 1
  The PEGS is designed for children with disabilities 5-9 years of age to indicate their perceived competence in performing 24 daily activities and to identify goals for therapy intervention. A higher score indicates higher perceived competence.

OTHER OUTCOMES:
Usability questionnaire | day 1
  The questionnaire is a 5-point Likert scale designed specifically for this study, a higher score indicating better user's perceptions on the usability.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Ju Kang, PhD, Principal Investigator — Chung Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided